CLINICAL TRIAL: NCT00075244
Title: A Phase I-II Pharmacokinetic/Pharmacodynamic Study of Replagal to Assess the Effects of Alternative Dose and Regimen in Patients With Fabry Disease
Brief Title: Alternative Dosing and Regimen of Replagal to Treat Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040073; 04-N-0073
Record Dates: First submitted 2004-01-06; First posted 2004-01-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Fabry Disease
Keywords: Lysosomes; Storage; Glycolipid; Fabry Disease; Stroke
MeSH Terms: conditions — Fabry Disease; Stroke | interventions — agalsidase alfa

INTERVENTIONS:
Drug: Replagal

SUMMARY:
The main goal of this study is to assess the pharmacodynamic effects of different or more frequent doses of Replagal compared to the standard dosing regimen. Replagal is a genetically engineered form of alpha-Galactosidase A, an enzyme that normally breaks down a fatty substance called globotriaosylceramide (Gb(3)). In patients with Fabry disease, GB(3) does not function properly and therefore builds up causing problems with the kidneys, heart, nerves, and blood vessels.

Male patients 18 years of age or older with Fabry disease who are not on dialysis and have not received a kidney transplant may be eligible for this study.

Participants are randomly assigned to receive one of the following five regimens of Replagal infusions, given through a vein over 20 to 80 minutes:

0.1 mg/kg body weight every week

0.2 mg/kg body weight every week

0.2 mg/kg body weight every other week

0.4 mg/kg body weight every week

0.4 mg/kg body wieght every other week

In the US, the infusions are given at the NIH Clinical Center. Vital signs are measured before, immediately after, and 1 hour after each infusion.

Baseline evaluations are done on an inpatient or outpatient basis. Baseline tests include a check of vital signs (temperature, respiratory rate, pulse rate, and blood pressure); physical examination; laboratory tests; and review of treatment side effects. Evaluations are also done at every infusion visit, and 1 week and 1 month after the last infusion.

Safety evaluations are done periodically and include vital sign measurements, physical examination, blood and urine tests, review of drug side effects, electrocardiogram (ECG), Holder monitor (2 hour ECG), and QSART (NIH only). The QSART (quantitative sudomotor axon reflex test) measures the amount of sweat in a particular area of skin, mostly the forearm. For this test, a cup partly filled with a liquid is strapped on the arm. A weak electric current is turned on, stimulating the sweat glands, and the amount of sweat produced is measured. There is a tingling sensation when the current is turned on.

Patients who complete the study will be offered the opportunity of receiving Replagal for 6 months in an extension study.

DETAILED DESCRIPTION:
OBJECTIVES: The goal of this study is to assess the pharmacodynamic effects of alternative weekly and every two week dosing regimens of Replagal (agalsidase alfa) in comparison to the current standard Replagal treatment regimen of 0.2 mg/kg given intravenously every two weeks.

STUDY POPULATION: Hemizygous males with Fabry disease who are 18 years of age or older.

DESIGN: This is a randomized, open-label study that will assess the pharmacodynamics and pharmacokinetics of five different dosing regimens of enzyme replacement therapy with Replagal. The effects of dose as well as dosing frequency will be evaluated and compared to the standard Replagal regimen.

OUTCOME MEASURES: The pharmacodynamic parameter to be assessed is plasma globotriaosylceramide (Gb3). The hypothesis to be tested is the role that frequency (weekly) and/or dose (0.1 to 0.4 mg/kg) of Replagal will play in pharmacodynamics as measured by reductions in plasma Gb3 compared to the current dose and frequency of 0.2 mg/kg given every two weeks. Clinical parameters including sweating, heart rate variability, proteinuria, severity of neuropathic pain, pain and anti-diarrheal medication usage, frequency and severity of abdominal pain, and frequency of diarrhea also will be assessed.

ELIGIBILITY:
INCLUSION CRITERIA:

Subject is a male hemizygote, age 18 years or older, with confirmed diagnosis of Fabry Disease. Diagnosis of Fabry disease may be confirmed by proof of a mutation of the alpha-Galactosidase A gene compatible with Fabry Disease and/or a deficiency of alpha-Galactosidase A (less than 4.0 nmol/mL/hour in plasma or serum or less than 8% of average mean normal in leukocytes).

Subject must have one or more clinical manifestations of Fabry disease including neuropathic pain, angiokeratoma, corneal verticillata, cardiomyopathy, hypo- or anhydrosis, abdominal pain and/or diarrhea, serum creatinine greater than 1.0 mg/dl or proteinuria greater than 300 mg/24 hours.

Subject must have voluntarily signed an Institutional Review Board (IRB) approved informed consent form after all relevant aspects of the study have been explained and discussed with the subject.

EXCLUSION CRITERIA:

Subject has been previously treated with Replagal or any other enzyme replacement therapy for Fabry Disease. If the patient has previously been treated with Replagal or another enzyme replacement therapy then they must have been off the therapy for at least 30 days and must have a Day-14 antibody blood sample drawn and that test must be negative for anti-agalsidase alfa IgG and IgE antibodies and not experienced a prior severe infusion reactions with prior enzyme replacement therapy.

Subject has been enrolled in another clinical investigative study in the past 30 days.

Subject is unable to give informed consent or is deemed unable to comply with all aspects of the clinical trial.

Subject has plasma Gb(3) drawn on Day -14 less than 4.0 nmol/mL.

Subject is undergoing dialysis or who has received a renal transplant.

Subjects who cannot tolerate the study procedures or who are unable or unwilling to travel to the study center as required by this protocol.

Subjects with an inter-current medical condition that would render them unsuitable for the study (e.g. HIV, diabetes) by confounding an assessment of the effects of the experimental therapy and its adverse events.

Subjects who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2004-01; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Brady RO, Gal AE, Bradley RM, Martensson E, Warshaw AL, Laster L. Enzymatic defect in Fabry's disease. Ceramidetrihexosidase deficiency. N Engl J Med. 1967 May 25;276(21):1163-7. doi: 10.1056/NEJM196705252762101. No abstract available. PMID 6023233
- [Background] Brady RO, Schiffmann R. Clinical features of and recent advances in therapy for Fabry disease. JAMA. 2000 Dec 6;284(21):2771-5. doi: 10.1001/jama.284.21.2771. PMID 11105184
- [Background] Meikle PJ, Hopwood JJ, Clague AE, Carey WF. Prevalence of lysosomal storage disorders. JAMA. 1999 Jan 20;281(3):249-54. doi: 10.1001/jama.281.3.249. PMID 9918480